CLINICAL TRIAL: NCT02753452
Title: Optimizing Life Success Through Residential Immersive Life Skills Programs for Youth With Disabilities
Brief Title: Optimizing Life Success Through Residential Immersive Life Skills (RILS) Programs for Youth With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: ErinoakKids Centre for Treatment and Development (Unknown); McMaster Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SSHRC-435-2014-0654; 14-506 (Other: Holland Bloorview Research Ethics Board)
Record Dates: First submitted 2016-04-08; First posted 2016-04-27 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Child-onset Disability
Keywords: youth; disability; transition; life skills; adolescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Residential Immersive Life Skills group (Active Comparator): Youth will take part in a residential life skills program of between one and three weeks, consisting of formal workshops, peer learning, outings in the community, one-on-one coaching and daily living tasks carried out with peers (e.g. cooking, laundry, grocery shopping).
  Interventions: Behavioral: Residential Immersive Life Skills programming
- Non-residential life skills program (Active Comparator): Youth will take part in programs focusing on increasing specific life skills, but taking place only during the day (i.e. non- residential).
  Interventions: Behavioral: Non-residential life skills programming
- Deferred RILS applicants (No Intervention): Youth who applied to a Residential Immersive Life Skills program but are deferred to a subsequent year. These youth are included as a comparator group to match the motivation level required to apply to a RILS program.
- No life skills program (No Intervention): Youth who did not apply or take part in any group life skills program. These youth provide a diagnosis and age matched comparator group.

INTERVENTIONS:
Behavioral: Residential Immersive Life Skills programming
  Arms: Residential Immersive Life Skills group
Behavioral: Non-residential life skills programming
  Arms: Non-residential life skills program

SUMMARY:
In Canada, between 3.6% and 7.7% of children under 19 years old are thought to have a chronic health condition that results in disability or limits to activity. These young people have difficulty finding jobs, attending school, living independently, and forming relationships with other people. These poorer life outcomes are partly the result of a lack of life skills. Life skills include the ability to solve problems and set goals, which allows youth to deal with the demands of everyday life. Several children's treatment centres in Ontario offer short-term residential immersive life skills (RILS) programs to provide youth with these life skills to help them take on adult roles. RILS programs are very promising in terms of making a long-term difference in youths' lives because they provide a place where youth can learn by doing, working with peers and taking risks in a safe environment. However, we do not yet know how well skills that are learned in RILS programs are kept up as time passes or how well RILS programs support broader skills, such as the ability to make one's own choices.

The proposed research will examine these issues and will ask the following questions:

1. What opportunities are youth given when they participate in RILS programs? What specific strategies do RILS service providers use to support youth in learning life skills?;
2. How do youth experience and perceive their participation in a RILS program, before, during and after they take part? What do their parents expect and experience in terms of their child's participation?; and
3. What changes do youth experience, particularly in terms of their ability to make choices for themselves and their sense of being able to cope with things that come up in their lives? The study will involve youth from several treatment centres in Ontario over the next three years.

Youth who are attending RILS programs will be compared with:

1. youth who are similar to the RILS youth, but who are taking part in a life skills program that is not residential;
2. youth who applied to a RILS program and were accepted, but who will take part in the program in a different year; and
3. a group of youth who are similar to the RILS youth but who are not taking part in any life skills program.

Youth will provide data at four time points: before the program starts, immediately after the program finishes, three months after the program is over and 12 months after the program is over.

ELIGIBILITY:
Inclusion Criteria:

* All youth must be between 14 and 21 years of age, have a child-onset disability, be able to set goals for themselves, and speak English.
* Parents who are enrolled must speak English.

Exclusion Criteria:

* Youth with severe behavioral issues will be excluded, since these would restrict the youth's ability to participate in a group learning experience.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Arc's Self-Determination Scale scores | Baseline, 1 week post intervention, 3 months post intervention, 12 months post intervention

SECONDARY OUTCOMES:
Change in General Self-Efficacy Scale scores | Baseline, 1 week post intervention, 3 months post intervention, 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gillian King, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Amy C McPherson, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McPherson AC, King G, Rudzik A, Kingsnorth S, Gorter JW; Ontario Independence Program Research (OIPR) team. Optimizing life success through residential immersive life skills programs for youth with disabilities: study protocol of a mixed-methods, prospective, comparative cohort study. BMC Pediatr. 2016 Sep 6;16(1):153. doi: 10.1186/s12887-016-0694-7. PMID 27600167